CLINICAL TRIAL: NCT03597113
Title: Growth and Compliance of Infants Fed an Extensively Hydrolyzed Hypo Allergenic Infant Formula
Brief Title: Evaluation of Infants Fed an Extensively Hydrolyzed Hypo Allergenic Infant Formula
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA16
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the growth and compliance of an intended use population of infants receiving an extensively hydrolyzed infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Infant is experiencing persistent feeding intolerance or allergy and diagnosed wtih Cow's Milk Protein Allergy (CMPA) or other condition where an extensively hydrolyzed formula is deemed appropriate by their healthcare professional
* Infants using OTC medications, home remedies, herbal preparations or rehydration fluids that might affect GI tolerance
* Parent(s) of infants enrolled on prescription medications, OTC medications, home remedies, herbal preparations or rehydration fluids directed by their healthcare professional, confirm their intention to continue their use during the study until directed by their healthcare professional to discontinue.
* Infant is not receiving steroids.
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* Parent(s) confirm their intention not to administer solid foods or juices to their infant from enrollment through the duration of the study
* Parent(s) confirm their intention not to administer vitamin or mineral supplements to their infant from enrollment through the duration of the study
* Infant's parent(s) or a LAR has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB)

Exclusion Criteria:

* Participation in another study that has not been approved as a concomitant study by AN

Ages: 0 Days to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be enrolled from outpatient clinics and physician offices.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline to Study Day 30
  Measured in Kg

SECONDARY OUTCOMES:
Formula Intake | Baseline to Study Day 30
  Parent completed diary

CONTACTS AND LOCATIONS:
Overall Officials: Aysugul Alptekin, MD, Study Chair — Abbott Turkey
Locations (46):
- Turkey (Türkiye) (46):
  - Adana City Hospital, Adana
  - Afyon Kocatepe University Medical Faculty, Afyonkarahisar
  - Ankara Dr. Sami Ulus Women and Child Disesase Research and Training Hospital B, Ankara
  - Hacettepe Üniversitesi University Medical Faculty A, Ankara
  - Hacettepe Üniversitesi University Medical Faculty B, Ankara
  - Ankara Dışkapı Child Disease Hospital A, Ankara
  - Ankara Dışkapı Child Disease Hospital B, Ankara
  - Ankara Research and Training Hospital, Ankara
  - Ankara Yıldırım Beyazıt University Yenimahalle Research and Training Hospital, Ankara
  - Gazi Üniversitesi University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty A, Antalya
  - Akdeniz University Medical Faculty B, Antalya
  - Balıkesir University Research and Training Hospital, Balıkesir
  - TC Sağlık Bilimleri University Bursa Yuksek Intisas Research and Training Hospital, Bursa
  - Pamukkale University Medical Faculty A, Denizli
  - Pamukkale University Medical Faculty B, Denizli
  - Fırat Üniversitesi University Medical Faculty, Elâzığ
  - Erzurum Research and Training Hospital, Erzurum
  - Gaziantep University Medical Faculty, Gaziantep
  - Hatay State Hospital, Hatay
  - İstanbul University İstanbul Medical School A, Istanbul
  - İstanbul University Cerrahpaşa Medical School, Istanbul
  - İstanbul Bakırköy Dr. Sadi Konuk Research and Training Hospital, Istanbul
  - Istanbul Esenler Women and Children Diseases Hospital, Istanbul
  - İstanbul Atakent Acıbadem Hospital, Istanbul
  - İstanbul Kanuni Sultan Süleyman Research and Training Hospital A, Istanbul
  - İstanbul Sisli Hamidiye Etfal Research and Training Hospital C, Istanbul
  - İstanbul Şişli Hamidiye Etfal Research and Training Hospital A, Istanbul
  - İstanbul Şişli Hamidiye Etfal Research and Training Hospital B, Istanbul
  - İstanbul Okmeydanı Research and Training Hospital, Istanbul
  - İstanbul Maslak Acıbadem Hospital, Istanbul
  - İstanbul Altunizade Acıbadem Hospital, Istanbul
  - İstanbul Göztepe Research and Training Hospital, Istanbul
  - İstanbul Ümraniye Research and Training Hospital A, Istanbul
  - İstanbul Ümraniye Research and Training Hospital B, Istanbul
  - Kocaeli Üniversitesi University Medical Faculty, Kocaeli
  - Konya Necmettin Erbakan University Medical Faculty, Konya
  - Konya Başkent University Hospital, Konya
  - Konya Selçuk University Medical Faculty, Konya
  - Kırıkkale University Medical Faculty, Kırıkkale
  - İnönü Üniversitesi University Medical Faculty, Malatya
  - Samsun Research and Training Hospital, Samsun
  - Karadeniz Teknik University Medical Faculty, Trabzon
  - Trabzon Kanuni Research and Training Hospital, Trabzon
  - Zonguldak Bülent Ecevit University Research and Training Hospital, Zonguldak

IPD SHARING:
Plan to Share IPD: Undecided